CLINICAL TRIAL: NCT05349357
Title: Compare the Effects of Sliding With Tensioner Technique of Neural Mobilization in Diabetic Peripheral Neuropathy Patients
Brief Title: Slider Versus Tensioner Neural Mobilization in Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC01253 Aaseya Syed
Record Dates: First submitted 2022-04-15; First posted 2022-04-27 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Diabetic Peripheral Neuropathic Pain
MeSH Terms: interventions — Muscle Stretching Exercises; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): TENS, Stretching exercises, ROM exercises Sliding neural mobilization to femoral, sciatic, tibial nerve
  Interventions: Other: Sliding Neural mobilization; Other: Stretching exercises; Device: TENS
- Group B (Active Comparator): TENS, Stretching exercises, ROM exercises Tensioner neural mobilization to femoral, sciatic, tibial nerve
  Interventions: Other: Tensioner Neural mobilization; Other: Stretching exercises; Device: TENS

INTERVENTIONS:
Other: Sliding Neural mobilization — Sliding neural mobilization to femoral, sciatic and tibial nerve
  Arms: Group A
Other: Tensioner Neural mobilization — Tensioner neural mobilization to femoral, sciatic and tibial nerve
  Arms: Group B
Other: Stretching exercises — Stretching exercises
Device: TENS — TENS

SUMMARY:
Neurodynamics, i.e., the mobilization of the peripheral nervous system, is a physical approach to the treatment of pain; the method relies on influencing pain physiology via mechanical treatment of neural tissues and the non-neural structures surrounding the nervous system. Neural mobilization (NM) is used to treat various disorders of the nervous system concerning the length and mobility of peripheral nerves, as the nerve mobilizing refers to techniques that help to reestablish motion between a nerve and its surrounding soft tissues, thus to treat the nerves that have become entangled within the soft tissue, as it leads to tension release on a nerve by stretching and pulling one end of the nerve during keeping the other end in a relaxed state.

DETAILED DESCRIPTION:
The neurodynamic technique both sliders and tensioners results in changes of the mechanical or physiological function of nerve tissues along with the interface; restoring pressure gradients, relieving hypoxia and pain resulting in reducing associated symptoms.

Through clinical reasoning the nervous system seems to be the logical place for treatment and explanations and previous descriptions of this method have clarified the overall impact on quality of life in diabetic peripheral neuropathy but it doesn't discuss which technique of neural mobilization is more effective and its effects on diabetic peripheral neuropathic population. Within this reasoning it is important to determine which neurodynamic technique is more effective in improving quality of life and reduce pain in patients with diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patient having≥12score on Self report Leads Assessment of Neuropathic Symptoms and Sign
* Patients with lower limb pain ≥4 to ≤7 on NPRS

Exclusion Criteria:

* Diabetic foot ulcer
* Complex regional pain syndrome
* Infection in lower limb
* Lower extremity amputation
* Discogenic pain
* Restricted joint deformity
* Dependency on chemical or drugs
* Pregnancy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-06-25 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Michigan neuropathy screening instrument | 3 weeks
  For screening the neuropathy; The MNSI questionnaire is self-administered. Responses are added to obtain a total score. 'Yes' responses to questions 1-3, 5-6, 8-9, 11-12, 14-15 are each counted as one point. 'No' responses to questions 7 and 13 each count as one point. Question 4 was considered to be a measure of impaired circulation and question 10 a measure of general asthenia and were not included in the published scoring algorithm. A score of ≥ 7 was considered abnormal. All 15 questions were included in the new scoring algorithms.
Numerical Pain Rating Scale | 3 weeks
  Quantify the pain ranging from 0 to 10 in which zero means no pain and 10 severe pain

SECONDARY OUTCOMES:
Quality of Life SF-36 | 3 weeks
  to assess the quality of life, SF-36 ; Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT(NMR), Principal Investigator — Riphah International University
Locations (1):
- DHQ Hospital, Mianwali, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pop-Busui R, Boulton AJ, Feldman EL, Bril V, Freeman R, Malik RA, Sosenko JM, Ziegler D. Diabetic Neuropathy: A Position Statement by the American Diabetes Association. Diabetes Care. 2017 Jan;40(1):136-154. doi: 10.2337/dc16-2042. No abstract available. PMID 27999003
- [Background] Iqbal Z, Azmi S, Yadav R, Ferdousi M, Kumar M, Cuthbertson DJ, Lim J, Malik RA, Alam U. Diabetic Peripheral Neuropathy: Epidemiology, Diagnosis, and Pharmacotherapy. Clin Ther. 2018 Jun;40(6):828-849. doi: 10.1016/j.clinthera.2018.04.001. Epub 2018 Apr 30. PMID 29709457
- [Background] Feldman EL, Nave KA, Jensen TS, Bennett DLH. New Horizons in Diabetic Neuropathy: Mechanisms, Bioenergetics, and Pain. Neuron. 2017 Mar 22;93(6):1296-1313. doi: 10.1016/j.neuron.2017.02.005. PMID 28334605
- [Background] Cho NH, Shaw JE, Karuranga S, Huang Y, da Rocha Fernandes JD, Ohlrogge AW, Malanda B. IDF Diabetes Atlas: Global estimates of diabetes prevalence for 2017 and projections for 2045. Diabetes Res Clin Pract. 2018 Apr;138:271-281. doi: 10.1016/j.diabres.2018.02.023. Epub 2018 Feb 26. PMID 29496507